CLINICAL TRIAL: NCT01110538
Title: The Massachusetts General Hospital Optical Coherence Tomography Registry
Status: Completed | Type: Observational
Sponsor: Ik-Kyung Jang, MD, PhD (Other)
Collaborators: Medtronic (Industry); Boston Scientific Corporation (Industry); Massachusetts General Hospital (Other)
Responsible Party: Sponsor-Investigator, Ik-Kyung Jang, MD, PhD, Professor of Medicine; Director, Cardiology Laboratory for Integrative Physiology & Imaging, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Other Study IDs: 2010-P-000387
Record Dates: First submitted 2010-04-22; First posted 2010-04-26 (Estimated); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Information will be collected prospectively in about 3,000 patients having Optical Coherence Tomography during cardiac catheterization. Subjects will be initially enrolled at sites outside of the United States, where Optical Coherence Tomography is approved by regulatory agencies. Subjects will be followed for up to 5 years.

DETAILED DESCRIPTION:
This project will create a prospective registry of 3,000 patients with follow-ups of up to 5 years.

The aims of the project will be:

1. identify plaque characteristics on OCT that are associated with adverse cardiac events including myocardial infarction
2. to identify characteristics of stented arteries that are associated with adverse events including restenosis and stent thrombosis

Because detailed clinical, angiographic and intravascular imaging data will be gathered from a large number of patients with clinical follow-ups, we anticipate that the registry will be a tremendous resource for additional research questions going forward.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have had OCT imaging performed during cardiac catheterization and have provided written consent

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who have intracoronary OCT imaging performed during cardiac catheterization are eligible for this registry. Subjects may be identified prior to or after cardiac catheterization and OCT imaging.
Sampling Method: Non-Probability Sample
Enrollment: 2714 (Actual)
Dates: Start 2010-08; Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiac events (MACE) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ik-Kyung Jang, M.D., Ph.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Seegers LM, Yeh DD, Wood MJ, Yonetsu T, Minami Y, Araki M, Nakajima A, Yuki H, Ako J, Soeda T, Kurihara O, Higuma T, Kimura S, Adriaenssens T, Nef HM, Lee H, McNulty I, Sugiyama T, Kakuta T, Jang IK. Cardiovascular Risk Factors and Culprit Plaque Characteristics in Women With Acute Coronary Syndromes. Am J Cardiol. 2023 Nov 15;207:13-20. doi: 10.1016/j.amjcard.2023.08.152. Epub 2023 Sep 16. PMID 37722196
- [Derived] Seegers LM, DeFaria Yeh D, Yonetsu T, Sugiyama T, Minami Y, Soeda T, Araki M, Nakajima A, Yuki H, Kinoshita D, Suzuki K, Niida T, Lee H, McNulty I, Nakamura S, Kakuta T, Fuster V, Jang IK. Sex Differences in Coronary Atherosclerotic Phenotype and Healing Pattern on Optical Coherence Tomography Imaging. Circ Cardiovasc Imaging. 2023 Aug;16(8):e015227. doi: 10.1161/CIRCIMAGING.123.015227. Epub 2023 Jul 28. PMID 37503629
- [Derived] Yuki H, Kinoshita D, Suzuki K, Niida T, Nakajima A, Seegers LM, Vergallo R, Fracassi F, Russo M, Di Vito L, Bryniarski K, McNulty I, Lee H, Kakuta T, Nakamura S, Jang IK. Layered plaque and plaque volume in patients with acute coronary syndromes. J Thromb Thrombolysis. 2023 Apr;55(3):432-438. doi: 10.1007/s11239-023-02788-9. Epub 2023 Mar 4. PMID 36869878
- [Derived] Seegers LM, Araki M, Nakajima A, Yonetsu T, Minami Y, Ako J, Soeda T, Kurihara O, Higuma T, Kimura S, Adriaenssens T, Nef HM, Lee H, McNulty I, Sugiyama T, Kakuta T, Jang IK. Sex Differences in Culprit Plaque Characteristics Among Different Age Groups in Patients With Acute Coronary Syndromes. Circ Cardiovasc Interv. 2022 Jun;15(6):e011612. doi: 10.1161/CIRCINTERVENTIONS.121.011612. Epub 2022 Jun 2. PMID 35652353
- [Derived] Nakajima A, Araki M, Kurihara O, Minami Y, Soeda T, Yonetsu T, Higuma T, Kakuta T, McNulty I, Lee H, Malhotra R, Nakamura S, Jang IK. Predictors for Rapid Progression of Coronary Calcification: An Optical Coherence Tomography Study. J Am Heart Assoc. 2021 Feb 2;10(3):e019235. doi: 10.1161/JAHA.120.019235. Epub 2021 Jan 26. PMID 33496191
- [Derived] Nakajima A, Minami Y, Araki M, Kurihara O, Soeda T, Yonetsu T, Wang Z, McNulty I, Lee H, Nakamura S, Jang IK. Optical Coherence Tomography Predictors for a Favorable Vascular Response to Statin Therapy. J Am Heart Assoc. 2021 Jan 5;10(1):e018205. doi: 10.1161/JAHA.120.018205. Epub 2020 Dec 19. PMID 33342228
- [Derived] Araki M, Yonetsu T, Kurihara O, Nakajima A, Lee H, Soeda T, Minami Y, McNulty I, Uemura S, Kakuta T, Jang IK. Predictors of Rapid Plaque Progression: An Optical Coherence Tomography Study. JACC Cardiovasc Imaging. 2021 Aug;14(8):1628-1638. doi: 10.1016/j.jcmg.2020.08.014. Epub 2020 Sep 30. PMID 33011121
- [Derived] Araki M, Soeda T, Kim HO, Thondapu V, Russo M, Kurihara O, Shinohara H, Minami Y, Higuma T, Lee H, Yonetsu T, Kakuta T, Jang IK. Spatial Distribution of Vulnerable Plaques: Comprehensive In Vivo Coronary Plaque Mapping. JACC Cardiovasc Imaging. 2020 Sep;13(9):1989-1999. doi: 10.1016/j.jcmg.2020.01.013. Epub 2020 Mar 16. PMID 32912472
- [Derived] Sugiyama T, Yamamoto E, Bryniarski K, Xing L, Fracassi F, Lee H, Jang IK. Coronary Plaque Characteristics in Patients With Diabetes Mellitus Who Presented With Acute Coronary Syndromes. J Am Heart Assoc. 2018 Jul 13;7(14):e009245. doi: 10.1161/JAHA.118.009245. PMID 30006490
- [Derived] Minami Y, Wang Z, Aguirre AD, Ong DS, Kim CJ, Uemura S, Soeda T, Lee H, Fujimoto J, Jang IK. Clinical Predictors for Lack of Favorable Vascular Response to Statin Therapy in Patients With Coronary Artery Disease: A Serial Optical Coherence Tomography Study. J Am Heart Assoc. 2017 Nov 1;6(11):e006241. doi: 10.1161/JAHA.117.006241. PMID 29092845
- [Derived] Yamamoto E, Siasos G, Zaromytidou M, Coskun AU, Xing L, Bryniarski K, Zanchin T, Sugiyama T, Lee H, Stone PH, Jang IK. Low Endothelial Shear Stress Predicts Evolution to High-Risk Coronary Plaque Phenotype in the Future: A Serial Optical Coherence Tomography and Computational Fluid Dynamics Study. Circ Cardiovasc Interv. 2017 Aug;10(8):e005455. doi: 10.1161/CIRCINTERVENTIONS.117.005455. PMID 28768758
- [Derived] Xing L, Higuma T, Wang Z, Aguirre AD, Mizuno K, Takano M, Dauerman HL, Park SJ, Jang Y, Kim CJ, Kim SJ, Choi SY, Itoh T, Uemura S, Lowe H, Walters DL, Barlis P, Lee S, Lerman A, Toma C, Tan JWC, Yamamoto E, Bryniarski K, Dai J, Zanchin T, Zhang S, Yu B, Lee H, Fujimoto J, Fuster V, Jang IK. Clinical Significance of Lipid-Rich Plaque Detected by Optical Coherence Tomography: A 4-Year Follow-Up Study. J Am Coll Cardiol. 2017 May 23;69(20):2502-2513. doi: 10.1016/j.jacc.2017.03.556. PMID 28521888
- [Derived] Ong DS, Lee JS, Soeda T, Higuma T, Minami Y, Wang Z, Lee H, Yokoyama H, Yokota T, Okumura K, Jang IK. Coronary Calcification and Plaque Vulnerability: An Optical Coherence Tomographic Study. Circ Cardiovasc Imaging. 2016 Jan;9(1):e003929. doi: 10.1161/CIRCIMAGING.115.003929. PMID 26743463
- [Derived] Vergallo R, Papafaklis MI, Yonetsu T, Bourantas CV, Andreou I, Wang Z, Fujimoto JG, McNulty I, Lee H, Biasucci LM, Crea F, Feldman CL, Michalis LK, Stone PH, Jang IK. Endothelial shear stress and coronary plaque characteristics in humans: combined frequency-domain optical coherence tomography and computational fluid dynamics study. Circ Cardiovasc Imaging. 2014 Nov;7(6):905-11. doi: 10.1161/CIRCIMAGING.114.001932. Epub 2014 Sep 4. PMID 25190591
- [Derived] Vergallo R, Joye R, Barlis P, Jia H, Tian J, Soeda T, Minami Y, Hu S, Dauerman HL, Toma C, Chan J, Lee H, Biasucci LM, Crea F, Jang IK. Bivalirudin versus unfractionated heparin for residual thrombus burden: a frequency-domain optical coherence tomography study. Catheter Cardiovasc Interv. 2015 Mar;85(4):575-82. doi: 10.1002/ccd.25631. Epub 2014 Aug 22. PMID 25115992
- [Derived] Jia H, Abtahian F, Aguirre AD, Lee S, Chia S, Lowe H, Kato K, Yonetsu T, Vergallo R, Hu S, Tian J, Lee H, Park SJ, Jang YS, Raffel OC, Mizuno K, Uemura S, Itoh T, Kakuta T, Choi SY, Dauerman HL, Prasad A, Toma C, McNulty I, Zhang S, Yu B, Fuster V, Narula J, Virmani R, Jang IK. In vivo diagnosis of plaque erosion and calcified nodule in patients with acute coronary syndrome by intravascular optical coherence tomography. J Am Coll Cardiol. 2013 Nov 5;62(19):1748-58. doi: 10.1016/j.jacc.2013.05.071. Epub 2013 Jun 27. PMID 23810884
- [Derived] Kato K, Yonetsu T, Jia H, Abtahian F, Vergallo R, Hu S, Tian J, Kim SJ, Lee H, McNulty I, Lee S, Uemura S, Jang Y, Park SJ, Mizuno K, Yu B, Jang IK. Nonculprit coronary plaque characteristics of chronic kidney disease. Circ Cardiovasc Imaging. 2013 May 1;6(3):448-56. doi: 10.1161/CIRCIMAGING.112.000165. Epub 2013 Mar 27. PMID 23536265